CLINICAL TRIAL: NCT02655133
Title: Effects on Sublingual Microcirculation of IgGAM Immunoglobulins (Pentaglobin®) in Severe Septic/Septic Shock Patients: a Randomized Controller Trial.
Brief Title: Effects on Microcirculation of IgGAM in Severe Septic/Septic Shock Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor of Anesthesiology, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgGAM-CLRZ-2014
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — pentaglobulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentaglobin® (Active Comparator): Patients will receive Immunoglobulins IgGAM (Pentaglobin®) at dosage of 250 mg/kg IV (5 mL/kg) per day (rate of 0.4 mL/kg/h), for 72 hours. Microcirculation will be monitored with sublingual microcirculation device (Cytocam®) and Near InfraRed Specrotcopy (NIRS, Hutchinson®).
  Interventions: Drug: Pentaglobin®
- Physiologic Solution (Placebo Comparator): Patients will receive physiologic solution (NaCl 0.9%) at a dosage of 5 ml/Kg per day for 72 hours. Microcirculation will be monitored with sublingual microcirculation device (Cytocam®) and Near InfraRed Specrotcopy (NIRS, Hutchinson®)
  Interventions: Drug: Physiologic solution

INTERVENTIONS:
Drug: Pentaglobin® — Immunoglobulins that will be used are IgM enriched and will be infused at 5 ml/Kg/day for 3 days.
  Other Names: IgGAM
  Arms: Pentaglobin®
Drug: Physiologic solution — Physiologic solution will be infused and will be infused at 5 ml/Kg/day for 3 days.
  Arms: Physiologic Solution

SUMMARY:
IgM-enriched immunoglobulins (IgGAM; Pentaglobin ® ) are new therapy for sepsis and septic shock since they support immune system especially in case of " immunoparalysis" . However IgGAM isn't commonly prescribed, few centres use it as routine in severe infections and there aren't any guidelines to determine how and when to use them.

Microcirculatory dysfunction is a crucial aspect in the pathogenesis of sepsis-induced organ dysfunction, resulting in hypoperfusion and tissue hypoxia. Unpublished clinical data suggest a beneficial effect of IgGAM at microvascular level proved with near infrared spectroscopy and Vascular occlusion test (VOT).

This study is a double blind phase II prospective randomised controlled trial that will include patients admitted to the Intensive Care Unit of the University Hospital "Ospedali Riuniti" of Ancona, after no more than 24 hours from development of severe sepsis or septic shoc.

Patients will be randomized into two groups (treaties and controls): patients in group of the treaties will be submitted to infusion of IgGAM conjugate (Pentaglobin ®) at dosage of 250 mg/kg IV (5 mL/kg) per day (rate of 0.4 mL/kg/h), for 72 hours. The controls will receive equal amount of physiological NaCl solution (0.9%) as placebo. Neither the patient nor the staff nurses and MD will be aware of the group and of the treatment applied. IgGAM solutions or NaCl 0.9% will be provided by the hospital pharmacy in similar bags. The remaining treatments will not be changed in any way and will be at the discretion of the doctor who's in charge of the patient. All patients of the two groups will receive the optimal therapy for their conditions, according to good medical clinical practice (GMP), with appropriate antibiotic therapy, vasoactive and infusional therapy

DETAILED DESCRIPTION:
Sepsis is a complex set of signs and symptoms caused by Systemic Inflammatory Response Syndrome (SIRS) to an infection. Sepsis-related mortality is directly proportional to the severity of organ dysfunction, and can be up to 80% in the case of septic shock.

Due to the pro-inflammatory response to this insult, tissues can be damaged far away from the primary site of infection. Concurrently with pro-inflammatory cytokines, the immune system produces anti-inflammatory mediators such as IL-10, which exert a compensatory antagonist response. The imbalance toward the anti-inflammatory one can conduce to "immuno-paralysis" that undermines the defense of the organism against infection.

Antibodies play a crucial role in fighting infections; low levels of protective antibodies are directly related to worst outcome. In consideration to that, polyvalent immunoglobulins (Ig) represent a potential therapeutic support for modulation of immune response and of inflammation in sepsis and septic shock.

They contain a broad spectrum of antibodies direct against a wide variety of bacterial antigens (all three classes normally found in human plasma - IgG and IgM and IgGAM conjugate).

In addition to antibody activity and antigen neutralization, benefits of Ig may include: inactivation of bacterial toxins (endotoxin and exotoxins); increased clearance of lipopolysaccharide; stimulation of leukocytes and their bactericidal activity through mechanism of opsonization; reduction in the activity of the classical pathway of the complement; modulation of cytokine production by blood mononuclear cells; synergistic activity with antibiotics.

Meta-analysis of main studies produced so far have shown that the Ig support, in particular the IgM-enriched ones, are associated with improved survival of patient with severe sepsis; these are promising results but the quality of the studies doesn't allow yet to have strong evidence in favour of their use.

The IgM-enriched immunoglobulins (IgGAM) proved to be most effective and are currently in the formulary and usable in case of severe infections (Pentaglobin ®). However, they are not commonly prescribed, and there aren't any guidelines to determine how and when to use them.

Unpublished clinical data suggest a beneficial effect even at microvascular level by application of the method of near infrared spectroscopy with vascular occlusion tests on level of tenar eminence of the hand.

Microcirculatory dysfunction (endothelial damage and glycocalyx, increased permeability and tissue edema, leukocyte adhesion, pro-coagulating agent, reduction of deformability of red blood cells) is a crucial aspect in the pathogenesis of sepsis-induced organ dysfunction, resulting in hypoperfusion and tissue hypoxia. Persistent microvascular perfusion abnormalities have been associated with an unfavorable outcome in patients with septic shock.

In consideration to that, a therapy that can prove to act on the microcirculation by restoring tissue perfusion would represent a promising pathophysiological approach to the patient in septic shock.

Material and Methods This is a double blind phase II prospective randomised controlled trial. It will include patients admitted to the Intensive Care Unit of the University Hospital "Ospedali Riuniti" of Ancona, after no more than 24 hours from development of severe sepsis or septic shock (diagnosis according to the criteria established by the Consensus Conference of 2001).

Patients younger than 18 years old, pregnant women, patients with severe sepsis/septic shock for more than 24 hours, chronic renal failure, terminal state with a life expectancy of less than 24 hours, contraindications to treatment with IgGAM, lack of informed consent will be excluded.

When inclusion criteria present and there aren't any exclusion criteria for this trials written informed consent will be taken by patient.

Demographic and clinical data will be collected by the investigator (age, weight, sex, acute and chronic diseases present at inclusion, GCS, APACHE II, SAPS II, arterial blood gases, SOFA score, lab data such as Hb, WBC, hepatic and renal function, blood sugar, Procalcitonin ) Patients will be randomized into two groups (treaties and controls): patients in Group of the treaties will be submitted to infusion of IgGAM conjugate (Pentaglobin ®) at dosage of 250 mg/kg IV (5 mL/kg) per day (rate of 0.4 mL/kg/h), for 72 hours. The controls will receive equal amount of physiological NaCl solution (0.9%) as placebo. Neither the patient nor the staff nurses and MD will be aware of the group and of the treatment applied (double blind trial). IgGAM solutions or NaCl 0.9% are provided by the hospital pharmacy in similar bags.

All patients of the two groups will receive the optimal therapy for their conditions, according to good medical clinical practice (GMP), with appropriate antibiotic therapy, vasoactive and infusional therapy.All treatments except from Pentaglobin/placebo will not be changed and will be at the discretion of the doctor who's in charge of the patient.At the time of inclusion, the following data will be collected: gender, age, anthropometric parameters, ICU admission diagnosis, known or suspected infection, results of microbiological tests. Prior to initiating therapy (T0), after 24 hours (T24) and at the end of therapy with IgGAM conjugate sublingual microcirculation will be evaluated by "Incident Dark Field Imaging (Medical imaging, Cytocam, IDF Braedius, Amsterdam, The Netherlands) and tissue oxygenation by using "Near Infrared Spectroscopy technique " (NIRS, InSpectra ™ Model 650; Hutchinson Technology Inc., Hutchinson, MN, USA). Both techniques are commonly used in our clinical practice and include CE mark.

At the same time points temperature and hemodynamic parameters (mean arterial pressure and heart rate; cardiac index, global end-diastolic volume, extravascular Lung water when monitored) will be collected, together with arterial and venous blood gas and lab data, diuresis and water balance, GCS. Concomitant treatments are noted. Data regarding the duration of hospital stay in intensive care and the outcome will be recorded.

The sample size has been assessed on the basis of the primary objective of the study, based on a significantly higher PVD in the Group of patients treated with IgGAM compared with controls at 72 hours after starting treatment. Assuming an average difference between the two groups at 72hrs of 4 mm/mm2 with a SD of 3, nine patients per group would be sufficient with an α error of 0.05 and a power of 80%. In total 20 patients will be included (10 per group All data will be collected anonymously, attributing to each selected patient only an alpha-numeric code, into an electronic database (password protected), respecting privacy and confidentiality of the data.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis
* septic shock

Exclusion Criteria:

* pregnant women
* severe sepsis/septic shock for more than 24 hours
* chronic renal failure
* terminal state with a life expectancy of less than 24 hours
* contraindications to treatment with IgGAM
* lack of informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Perfused vessel density (PVD) | 72 hours
  The perfused vessel density (PVD), unity of measure mm/mm2, is detected in vivo by Incident Dark Field Imaging at sublingual microcirculation. It represents the quantity of well perfused vessels at microcirculatory level.

SECONDARY OUTCOMES:
StO2 upload | 72 hours
  StO2 upslope (%/min) is measured with Near InfraRed Spectroscopy at the tenar muscle. It represents the velocity of the recovery of the tissue oxygen saturation after a short period of ischemia of the hand, the Vascular Occlusion Test.
Microcirculatory Flow Index (MFI) | 72 hours
  Microcirculatory Flow Index detected in vivo by Incident Dark Field Imaging at sublingual microcirculation. It represents the quality of blood flow at microcirculatory level.
Arterial blood lactate | 72 hours
  It represents the level of anaerobic metabolism of the body
SOFA score (Sequential Organ Failure Assessment) | 72 hours
  It represents the organ dysfuntion/failure of each patients

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, Principal Investigator — AOU Ospedali Riuniti di Ancona, Italy
Locations (1):
- University ICU, AOU Ospedali Riuniti Ancona, Torrette Di Ancona, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domizi R, Adrario E, Damiani E, Scorcella C, Carsetti A, Giaccaglia P, Casarotta E, Gabbanelli V, Pantanetti S, Lamura E, Ciucani S, Donati A. IgM-enriched immunoglobulins (Pentaglobin) may improve the microcirculation in sepsis: a pilot randomized trial. Ann Intensive Care. 2019 Dec 3;9(1):135. doi: 10.1186/s13613-019-0609-5. PMID 31797105